CLINICAL TRIAL: NCT00066573
Title: A Randomized Phase III Trial Of Exemestane Versus Anastrozole In Postmenopausal Women With Receptor Positive Primary Breast Cancer
Brief Title: Exemestane or Anastrozole in Treating Postmenopausal Women Who Have Undergone Surgery for Primary Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network); ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA27; CAN-NCIC-MA27 (Other: Cancer.gov); NCCTG-MA27 (Other: NCCTG); CALGB-CAN-NCIC-MA27 (Other: CALGB); ECOG-CAN-NCIC-MA27 (Other: ECOG); SWOG-CAN-NCIC-MA27 (Other: SWOG); IBCSG-30-04 (Other: IBCSG); 2005-001893-28 (EudraCT Number); CDR0000316325 (Other: PDQ); NCT00438529 (obsolete NCT alias)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exemestane (Experimental): Patients receive oral exemestane (25 mg) once daily for 5 years.
  Interventions: Drug: exemestane
- Anastrozole (Active Comparator): Patients receive oral anastrozole (1 mg) once daily for 5 years.
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: anastrozole — Given orally
  Arms: Anastrozole
Drug: exemestane — Given orally
  Arms: Exemestane

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy, using exemestane or anastrozole, may fight breast cancer by reducing the production of estrogen. It is not yet known whether exemestane is more effective than anastrozole in preventing the recurrence of breast cancer.

PURPOSE: This randomized phase III trial is studying exemestane to see how well it works compared to anastrozole in preventing cancer recurrence in postmenopausal women who have undergone surgery for primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free survival of postmenopausal women with receptor-positive primary breast cancer when treated with exemestane vs anastrozole.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the time to distant recurrence in patients treated with these regimens.
* Compare the incidence of new primary contralateral breast cancer in patients treated with these regimens.
* Compare the incidence of all clinical fractures, specifically hip and vertebral fractures, in patients treated with these regimens.
* Compare cardiovascular morbidity and mortality (i.e., significant coronary heart disease, which includes myocardial infarctions and angina requiring percutaneous transluminal coronary angioplasty or coronary artery bypass graft, fatal and nonfatal strokes, and all vascular deaths) in patients treated with these regimens.
* Correlate therapy induced changes in breast density with plasma hormones and growth factors, drug levels of exemestane and anastrozole, genetic variation and breast cancer recurrence or contralateral events in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to lymph node status at diagnosis (negative vs positive vs unknown), prior adjuvant chemotherapy (yes vs no), and herceptin use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral exemestane (25 mg) once daily for 5 years.
* Arm II: Patients receive oral anastrozole (1 mg) once daily for 5 years. In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months during the first year of study participation and annually thereafter.

PROJECTED ACCRUAL: A total of 6,840 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * pT1-3; pNX, pN0-2 or pN3*; M0
  * Neoadjuvant patients are eligible no earlier than 3 weeks or later than 3 months after excisional surgery, provided both the clinical-diagnostic staging of cancer and postsurgical resection-pathologic staging of cancer meet the requirements for primary tumor, regional lymph nodes, and distant metastasis classification NOTE: *Only when the sole basis for this classification is the presence of 10 or more involved axillary lymph nodes
* Completely resected disease

  * Primary surgery performed at least 3 weeks but no more than 3 months before study entry (if no chemotherapy was given)

    * Primary surgery is defined as the last surgery at which histologic evidence of invasive or in situ disease was present in the pathology specimen
  * Patients with positive sentinel lymph node biopsy are eligible provided they have had a subsequent axillary lymph node dissection
* No metachronous breast cancer
* Bilateral mammogram within the past 12 months unless initial surgery was a total mastectomy, in which case only a mammogram of the remaining breast is required
* No metastases confirmed by 1 of the following methods:

  * Bone scan* (required only if alkaline phosphatase is at least 2 times normal and/or there are symptoms of metastatic disease)
  * Abdominal ultrasound or CT scan (required only if AST/ALT or alkaline phosphatase is at least 2 times normal, unless the elevation is in the bone fraction)
  * Chest x-ray NOTE: *Confirmatory x-ray, CT scan, or MRI required if the bone scan results are questionable
* No locally recurrent disease
* No prior or concurrent carcinoma in situ of the contralateral breast treated with partial mastectomy and/or hormonal therapy

  * Patients with prior or concurrent carcinoma in situ of the ipsilateral breast are eligible provided the tumor was completely excised AND they have not received prior hormonal therapy
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive by immunohistochemistry or tumor receptor content ≥ 10 fmol/mg protein

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal prior to chemotherapy, defined as 1 of the following:

  * Over 60 years of age
  * Age 45-59 with spontaneous cessation of menses for more than 1 year prior to study entry
  * Age 45-59 with menses ceasing (secondary to hysterectomy or spontaneously) within the past year AND a follicle-stimulating hormone (FSH) level prior to study entry in the postmenopausal range*
  * Age 45-59, previously on hormone replacement therapy (HRT) and have discontinued HRT upon diagnosis of this malignancy AND has an FSH level prior to study entry in the postmenopausal range*
  * Has undergone bilateral oophorectomy NOTE: *By institutional standards OR > 34.4 IU/L if institutional range is not available)

Performance status

* ECOG 0-2

Life expectancy

* At least 5 years

Hematopoietic

* WBC at least 3,000/mm^3 OR
* Granulocyte count at least 1,500/mm^3 AND
* Platelet count at least 100,000/mm^3

Hepatic

* See Disease Characteristics
* AST and/or ALT less than 2 times upper limit of normal (ULN)*
* Alkaline phosphatase less than 2 times ULN* NOTE: *Unless imaging examinations have ruled out metastatic disease

Renal

* Not specified

Other

* Able to swallow study medication and have adequate unassisted oral intake in order to maintain reasonable nutrition status
* No other non-breast malignancy within the past 5 years except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid tumors with no evidence of disease for at least 5 years
* No other concurrent medical or psychiatric condition that would preclude study participation and/or interfere with results

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior and concurrent trastuzumab (Herceptin®) allowed

Chemotherapy

* See Disease Characteristics
* At least 3 weeks but no more than 3 months since prior chemotherapy
* Prior adjuvant chemotherapy allowed

Endocrine therapy

* See Disease Characteristics
* No prior aromatase inhibitor
* No prior tamoxifen or other selective estrogen receptor modulators (SERMs) except raloxifene

  * At least 3 weeks since prior raloxifene
* At least 3 weeks since prior and no concurrent over-the-counter products or supplements considered to have an estrogenic effect, including any of the following:

  * Ginseng
  * Ginkgo biloba
  * Black cohosh
  * Dong quai
  * Fortified soy supplements (e.g., phytoestrogen preparations)
* At least 3 weeks since other prior hormonal therapy or steroids considered to have an estrogenic effect
* No concurrent estrogens, progesterones, androgens, or SERMs

  * Concurrent intermittent vaginal estrogens (e.g., vagifem, estrogen vaginal cream, testosterone, estradiol vaginal gel, or Estring) allowed if other local measures for intractable vaginal atrophy are insufficient
* No other concurrent therapy that would have an estrogenic effect, including endocrine therapy, hormonal therapy, or steroid therapy

Radiotherapy

* See Disease Characteristics
* Prior adjuvant radiotherapy allowed
* Concurrent radiotherapy allowed

Surgery

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7576 (Actual)
Dates: Start 2003-06-06 (Actual); Primary Completion 2010-11-07 (Actual); Study Completion 2012-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital; James N. Ingle, MD, Study Chair — Mayo Clinic; Matthew J. Ellis, MD, PhD, FRCP, Study Chair — Washington University Siteman Cancer Center; George W. Sledge, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center; George T. Budd, MD, Study Chair — The Cleveland Clinic; Manuela Rabaglio, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (39):
- Canada (39):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Lethbridge Cancer Centre, Lethbridge, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Quinte Healthcare Corporation, Belleville, Ontario
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Regional Cancer Program of the Hopital Regional, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Centre - West Toronto, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Centre de Sante et de services sociaux de Gatineau, Gatineau, Quebec
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moy B, Elliott CR, Chapman J-AW, et al.: NCIC CTG MA.27: menopausal symptoms of ethnic minority women. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-3059, S144, 2006.
- [Result] Goss PE, Ingle JN, Pritchard KI, Ellis MJ, Sledge GW, Budd GT, Rabaglio M, Ansari RH, Johnson DB, Tozer R, D'Souza DP, Chalchal H, Spadafora S, Stearns V, Perez EA, Liedke PE, Lang I, Elliott C, Gelmon KA, Chapman JA, Shepherd LE. Exemestane versus anastrozole in postmenopausal women with early breast cancer: NCIC CTG MA.27--a randomized controlled phase III trial. J Clin Oncol. 2013 Apr 10;31(11):1398-404. doi: 10.1200/JCO.2012.44.7805. Epub 2013 Jan 28. PMID 23358971
- [Derived] Chapman JW, Bayani J, SenGupta S, Bartlett JMS, Piper T, Quintayo MA, Virk S, Goss PE, Ingle JN, Ellis MJ, Sledge GW, Budd GT, Rabaglio M, Ansari RH, Tozer R, D'Souza DP, Chalchal H, Spadafora S, Stearns V, Perez EA, Gelmon KA, Whelan TJ, Elliott C, Shepherd LE, Chen BE, Taylor KJ. Adjunctive Statistical Standardization of Adjuvant Estrogen Receptor and Progesterone Receptor in Canadian Cancer Trials Group MA.27 Postmenopausal Breast Cancer Trial of Exemestane Versus Anastrozole. J Clin Oncol. 2024 Aug 20;42(24):2887-2898. doi: 10.1200/JCO.24.00835. Epub 2024 Jun 2. PMID 38824432
- [Derived] Ethier JL, Anderson GM, Austin PC, Clemons M, Parulekar W, Shepherd L, Summers Trasiewicz L, Tu D, Amir E. Influence of the competing risk of death on estimates of disease recurrence in trials of adjuvant endocrine therapy for early-stage breast cancer: A secondary analysis of MA.27, MA.17 and MA.17R. Eur J Cancer. 2021 May;149:117-127. doi: 10.1016/j.ejca.2021.02.034. Epub 2021 Apr 11. PMID 33853037
- [Derived] Strasser-Weippl K, Higgins MJ, Chapman JW, Ingle JN, Sledge GW, Budd GT, Ellis MJ, Pritchard KI, Clemons MJ, Badovinac-Crnjevic T, Han L, Gelmon KA, Rabaglio M, Elliott C, Shepherd LE, Goss PE. Effects of Celecoxib and Low-dose Aspirin on Outcomes in Adjuvant Aromatase Inhibitor-Treated Patients: CCTG MA.27. J Natl Cancer Inst. 2018 Sep 1;110(9):1003-1008. doi: 10.1093/jnci/djy017. PMID 29554282
- [Derived] Strasser-Weippl K, Sudan G, Ramjeesingh R, Shepherd LE, O'Shaughnessy J, Parulekar WR, Liedke PER, Chen BE, Goss PE. Outcomes in women with invasive ductal or invasive lobular early stage breast cancer treated with anastrozole or exemestane in CCTG (NCIC CTG) MA.27. Eur J Cancer. 2018 Feb;90:19-25. doi: 10.1016/j.ejca.2017.11.014. Epub 2017 Dec 20. PMID 29274617
- [Derived] Yerushalmi R, Dong B, Chapman JW, Goss PE, Pollak MN, Burnell MJ, Levine MN, Bramwell VHC, Pritchard KI, Whelan TJ, Ingle JN, Shepherd LE, Parulekar WR, Han L, Ding K, Gelmon KA. Impact of baseline BMI and weight change in CCTG adjuvant breast cancer trials. Ann Oncol. 2017 Jul 1;28(7):1560-1568. doi: 10.1093/annonc/mdx152. PMID 28379421
- [Derived] Stearns V, Chapman JA, Ma CX, Ellis MJ, Ingle JN, Pritchard KI, Budd GT, Rabaglio M, Sledge GW, Le Maitre A, Kundapur J, Liedke PE, Shepherd LE, Goss PE. Treatment-associated musculoskeletal and vasomotor symptoms and relapse-free survival in the NCIC CTG MA.27 adjuvant breast cancer aromatase inhibitor trial. J Clin Oncol. 2015 Jan 20;33(3):265-71. doi: 10.1200/JCO.2014.57.6926. Epub 2014 Dec 15. PMID 25512454
- [Derived] Goetz MP, Schaid DJ, Wickerham DL, Safgren S, Mushiroda T, Kubo M, Batzler A, Costantino JP, Vogel VG, Paik S, Carlson EE, Flockhart DA, Wolmark N, Nakamura Y, Weinshilboum RM, Ingle JN, Ames MM. Evaluation of CYP2D6 and efficacy of tamoxifen and raloxifene in women treated for breast cancer chemoprevention: results from the NSABP P1 and P2 clinical trials. Clin Cancer Res. 2011 Nov 1;17(21):6944-51. doi: 10.1158/1078-0432.CCR-11-0860. Epub 2011 Aug 31. PMID 21880792

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exemestane | Anastrozole
Started | 3789 | 3787
Completed | 3761 | 3759
Not Completed | 28 | 28
Not completed — Did not received protocol treatment | 28 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane | Anastrozole | Total
Number analyzed (Participants) | 3789 | 3787 | 7576
Age, Continuous [Median (Full Range); unit: years] | 63.9 [35.9 to 93.6] | 64.3 [32.3 to 95.1] | 64.1 [32.3 to 95.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3789 | 3787 | 7576
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event free survival, the primary endpoint of this study, is defined as the time from randomization to the time of documented locoregional or distant recurrence, new primary breast cancer, or death from any cause.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 3789 | 3787
percentage of participants | 88 [87 to 89] | 89 [88 to 90]
Statistical Analysis 1: Comparison: Exemestane vs Anastrozole; Test type: Superiority — To detect a hazard ratio (HR) of 0.80 between exemestane and anastrozole (ie, an improvement in 5-year EFS from 87.5% to 89.9%, with a two-sided 5% level test and 80% power, 6,840 patients and 630 events were needed for final analysis; p = 0.85, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.87 to 1.18]

2. Secondary Outcome: Overall Survival: Percentage of Participants Alive at 5 Years
Description: Overall survival is defined as the time from randomization to the time of death from any cause.
Time Frame: 5 years
Population: Intend to treat
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 3789 | 3787
Percentage of Participants | 92 [91 to 93] | 92 [91 to 93]
Statistical Analysis 1: Comparison: Exemestane vs Anastrozole; Test type: Superiority — No power calculation for secondary analysis; p = 0.46, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.77 to 1.13]

3. Secondary Outcome: Distant Disease-free Survival: Number of Participants Without Documented Distant Recurrence
Description: Time to distant disease-free survival (DDFS) is defined as the time from randomization to the time of documented distant recurrence. Distant recurrence is the cancer coming back in a part of the body away from the breast, such as the bones or liver.
Time Frame: 5 years
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 3789 | 3787
Participants | 157 | 164

4. Secondary Outcome: Clinical Fracture Rate: Number of Participants With Bone Fractures.
Description: Clinical fracture at any time, including hip, spine, wrist fractures and other bone fractures.
Time Frame: 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane | Anastrozole
Number analyzed (Participants) | 3789 | 3787
Participants | 358 | 354

ADVERSE EVENTS:
Time Frame: 8 years
Description: Participants at Risk of Adverse Event or SAE were those who received at least one dose of protocol therapy.
Arm/Group | Exemestane | Anastrozole
Serious Adverse Events (participants affected / at risk) | 19/3761 | 7/3759
Other Adverse Events (participants affected / at risk) | 3556/3761 | 3543/3759
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=3761) | Anastrozole (N=3759)
Cardiac ischemia/infarction (Cardiac disorders) | 3 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Supraven.arrhyth. Atrial flutter (Cardiac disorders) | 1 | 0
Ventric.arrhyth. Trigeminy (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Nyctalopia (Eye disorders) | 0 | 1
Ocular - Other (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Bilirubin (Investigations) | 1 | 0
Creatinine (Investigations) | 1 | 0
cTnI (Investigations) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
CNS ischemia (Nervous system disorders) | 3 | 1
Neurology - Other (Nervous system disorders) | 1 | 0
Neuropathy-motor (Nervous system disorders) | 0 | 1
Neuropathy: cranial CN VIII (Nervous system disorders) | 1 | 0
Speech impairment (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 1 | 0
Incontinence, urinary (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=3761) | Anastrozole (N=3759)
Constipation (Gastrointestinal disorders) | 614 | 606
Diarrhea (Gastrointestinal disorders) | 464 | 414
Flatulence (Gastrointestinal disorders) | 399 | 363
Heartburn (Gastrointestinal disorders) | 574 | 556
Nausea (Gastrointestinal disorders) | 436 | 442
Pain Abdomen NOS (Gastrointestinal disorders) | 202 | 220
Edema: limb (General disorders) | 749 | 760
Fatigue (General disorders) | 1697 | 1749
Fracture (Injury, poisoning and procedural complications) | 290 | 292
Cholesterol (Investigations) | 591 | 677
Weight gain (Investigations) | 257 | 286
Weight loss (Investigations) | 229 | 218
Anorexia (Metabolism and nutrition disorders) | 238 | 249
Hyperglycemia (Metabolism and nutrition disorders) | 347 | 373
Arthritis (Musculoskeletal and connective tissue disorders) | 264 | 242
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1243 | 1369
Pain Back (Musculoskeletal and connective tissue disorders) | 480 | 504
Pain Bone (Musculoskeletal and connective tissue disorders) | 381 | 410
Pain Extremity-limb (Musculoskeletal and connective tissue disorders) | 468 | 511
Pain Joint (Musculoskeletal and connective tissue disorders) | 2085 | 2086
Pain Muscle (Musculoskeletal and connective tissue disorders) | 667 | 629
Dizziness (Nervous system disorders) | 526 | 504
Neuropathy-sensory (Nervous system disorders) | 576 | 528
Pain Head/headache (Nervous system disorders) | 414 | 399
Insomnia (Psychiatric disorders) | 574 | 521
Mood alteration Anxiety (Psychiatric disorders) | 258 | 229
Mood alteration Depression (Psychiatric disorders) | 374 | 377
Pain Breast (Reproductive system and breast disorders) | 288 | 312
Vaginal dryness (Reproductive system and breast disorders) | 248 | 260
Cough (Respiratory, thoracic and mediastinal disorders) | 671 | 666
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 656 | 652
Alopecia (Skin and subcutaneous tissue disorders) | 235 | 212
Rash (Skin and subcutaneous tissue disorders) | 474 | 437
Sweating (Skin and subcutaneous tissue disorders) | 626 | 603
Hot flashes (Vascular disorders) | 2086 | 2138
Hypertension (Vascular disorders) | 300 | 326

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes